CLINICAL TRIAL: NCT04523532
Title: Effect of Intervention With Dietary Folate and Hazelnut Oil on the Methylation Levels of the LEP and POMC Genes, Body Weight and Lipid Profile of Overweight Women
Brief Title: Dietary Intervention and Assessment of Obesity-related Gene Methylation Levels in Overweight Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thamires Ribeiro Chaves (Other)
Responsible Party: Sponsor-Investigator, Thamires Ribeiro Chaves, Principal Investigator, Federal University of Paraíba
Organization: Federal University of Paraíba (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TChaves
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-08

CONDITIONS: Obesity
Keywords: Epigenetic; Obesity; Diet; Folate; Monounsaturated fat
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Folate + hazelnut oil (Experimental): Group 1 = in this group, the individuals received, during the period of 08 weeks daily, daily dietary intervention with, 300 g of vegetables rich in folate - 191µg and additionally received 01 capsule containing 25 mg hazelnut oil per day.
  Interventions: Other: Dietary folate and hazelnut oil
- Group 2: Folate (Placebo Comparator): Group 2 = in this group, the individuals received, during the period of 08 weeks daily, daily dietary intervention with, 300 g of folate-rich vegetables - 191 µg and 01 placebo capsule.
  Interventions: Other: Dietary folate and hazelnut oil
- Group 3: Moderate folate + hazelnut oil (Experimental): Group 3 = in this group, individuals received, during the period of 08 weeks daily, with 300 g of vegetables containing 94 µg of folate and 01 capsule containing 25 mg of hazelnut oil per day.
  Interventions: Other: Dietary folate and hazelnut oil
- Group 4: Control (No Intervention): Group 4 = in this group, individuals received weekly visits during the 08 week period to maintain their eating habits.

INTERVENTIONS:
Other: Dietary folate and hazelnut oil — Intervention with folate-rich diet and hazelnut oil supplement in capsule
  Arms: Group 1: Folate + hazelnut oil; Group 2: Folate; Group 3: Moderate folate + hazelnut oil

SUMMARY:
The clinical study aimed to study the effect of an intervention with foods containing folate and hazelnut oil to assess whether this diet could modulate the methylation levels of two obesity-related genes, LEP and POMC, in addition to impacting body weight and values of lipid profile of overweight women. The hypothesis of the clinical study is that the intervention diet could reduce the methylation levels of the genes mentioned and this would impact on the reduction of body weight and improvement of the lipid profile of the women studied.

DETAILED DESCRIPTION:
The intervention study was carried out with a sample selected by randomization, and n = 40 adult women classified as overweight were considered for the study. After assessing the eligibility criteria, women were instructed to have stable weight, eating habits and levels of physical activity constant to those found during the baseline, as well as receiving an individual diet plan one week before starting the dietary intervention. Before the start of the intervention, the 40 women were allocated to four groups of 10 each, and three groups started the individual diet plan for weight maintenance with a focus on vegetables and legumes with antioxidant and folate-rich action, and were also invited to consume foods fortified with folic acid and foods naturally rich in folate to achieve a usual folate intake close to the RAS (≥400 µg), this amount was for intervention group 1 and 2, group 3 received a lower amount (approximately half of the consumption of groups 1 and 2) and group 4 was the control group.

Still referring to the intervention, the participants of the three groups received advice from a nutritionist, responsible for this research and all the printed material free of charge, including pre-packaged foods, and also delivered hazelnut oil capsules, used as a source of monounsaturated fat. Counseling sessions with the nutritionist were offered daily at the homes during the entire period of the intervention, except for group 4, where the monitoring was weekly, to maintain eating habits.

After the end of the 8 weeks of the intervention, the third stage of the study began, which consisted of anthropometric assessment, analysis of the dietary intake of the 24-hour food record and blood collection for biochemical tests and DNA methylation.

ELIGIBILITY:
Inclusion Criteria:

* Adult women, aged between 20 and 59 years;
* Women with classification of overweight and obesity;
* Women who signed the informed consent form.

Exclusion Criteria:

* Women who changed their lifestyle 3 months before the study started;
* Alcoholic women or smokers;
* Taking medications known to interfere with folic acid metabolism (in the past 3 months), such as antacids and anticonvulsants;
* Individuals who use supplements in general, such as fish oil or other fatty acids;
* Pregnant or planning to become pregnant during the study period.

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
DNA methylation levels | week 8
  For analysis of methylation levels the blood of the participants was collected, chosen for analysis, as it is a metabolically active tissue, with an important role in the adverse inflammatory and vascular consequences of adiposity, being widely used for the purpose of clinical diagnosis

SECONDARY OUTCOMES:
Food intake | week 8
  It is a method that describes a wide variety of foods, Reminder 24h (R24h) is used when you want to compare the average nutrient intake of different populations.

OTHER OUTCOMES:
Folate food intake | week 8
  Three 24-hour reminders were used to assess folate intake, subsequently analyzed in food software and to estimate habitual consumption and correct intrapersonal variance, the online multi-source method (MSM), available on the website, (https: // msm .dife.de / tps / msm /). MSM is a statistical technique proposed by the European Prospective Investigation into cancer and Nutrition.
Oleic Acid food intake | week 8
  Three 24-hour reminders were used to assess oleic acid intake, subsequently analyzed in food software and to estimate habitual consumption and correct intrapersonal variance, the online multi-source method (MSM), available on the website, (https: // msm .dife.de / tps / msm /). MSM is a statistical technique proposed by the European Prospective Investigation into cancer and Nutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Lima, Study Director — Federal University of Paraíba
Locations (1):
- Raquel Patrícia Ataíde Lima, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Sociodemographic data, food consumption, anthropometric assessment, biochemical tests and DNA methylation of the participants. And all the statistical data that support the study.
Supporting Information: Study Protocol, SAP
Time Frame: 30 days after publication
Access Criteria: Online access to researchers

REFERENCES:
- [Result] Lima RPA, do Nascimento RAF, Luna RCP, Persuhn DC, da Silva AS, da Conceicao Rodrigues Goncalves M, de Almeida ATC, de Moraes RM, Junior EV, Fouilloux-Meugnier E, Vidal H, Pirola L, Magnani M, de Oliveira NFP, Prada PO, de Carvalho Costa MJ. Effect of a diet containing folate and hazelnut oil capsule on the methylation level of the ADRB3 gene, lipid profile and oxidative stress in overweight or obese women. Clin Epigenetics. 2017 Oct 13;9:110. doi: 10.1186/s13148-017-0407-6. eCollection 2017. PMID 29046732
- Available data/document: Study Protocol — http://clinicalepigeneticsjournal.biomedcentral.com/articles/10.1186/s13148-017-0407-6